CLINICAL TRIAL: NCT04590586
Title: Industry Alliance Platform Trial to Assess the Efficacy and Safety of Multiple Candidate Agents for the Treatment of COVID-19 in Hospitalized Patients
Brief Title: Study of Multiple Candidate Agents for the Treatment of COVID-19 in Hospitalized Patients
Acronym: COMMUNITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COV-01
Record Dates: First submitted 2020-10-14; First posted 2020-10-19 (Actual); Results first posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Severe acute respiratory syndrome coronavirus 2
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care; apremilast; lanadelumab; zilucoplan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Apremilast + Standard of Care (Experimental): Participants will be randomized to receive 30 mg apremilast orally twice a day (BID) in addition to standard of care treatment for 14 days or until hospital discharge, death, or discontinuation of investigational product, whichever occurred first.
  Interventions: Drug: Standard of care; Drug: Apremilast
- Apremilast Placebo + Standard of Care (Placebo Comparator): Participants will be randomized to receive matching placebo to apremilast orally twice a day in addition to standard of care treatment for 14 days or until hospital discharge, death, or discontinuation of investigational product, whichever occurred first.
  Interventions: Drug: Standard of care; Drug: Apremilast placebo
- Lanadelumab + Standard of Care (Experimental): Participants will be randomized to receive lanadelumab 300 mg by intravenous infusion on Day 1, and a second dose administered on Day 4 in addition to standard of care.
  Interventions: Drug: Standard of care; Drug: Lanadelumab
- Lanadelumab Placebo + Standard of Care (Placebo Comparator): Participants will be randomized to receive placebo to lanadelumab by intravenous infusion on Day 1, and a second dose administered on Day 4 in addition to standard of care.
  Interventions: Drug: Standard of care; Drug: Lanadelumab placebo
- Zilucoplan + Standard of Care (Experimental): Participants will be randomized to receive 32.4 mg zilucoplan by subcutaneous injection every day for 14 days, or until discharge if discharge was before 14 days of treatment in addition to standard of care.
  Interventions: Drug: Standard of care; Drug: Zilucoplan
- Zilucoplan Placebo + Standard of Care (Placebo Comparator): Participants will be randomized to receive placebo to zilucoplan by subcutaneous injection every day for 14 days, or until discharge if discharge was before 14 days of treatment in addition to standard of care.
  Interventions: Drug: Standard of care; Drug: Zilucoplan placebo

INTERVENTIONS:
Drug: Standard of care — Standard of care (SoC) treatment for COVID-19 infection in line with institutional practice. The SoC may change as new information becomes available about treating COVID-19.
Drug: Apremilast — Apremilast administered orally as a tablet.
  Other Names: Otezla
  Arms: Apremilast + Standard of Care
Drug: Apremilast placebo — Matching apremilast placebo administered orally as a tablet.
  Arms: Apremilast Placebo + Standard of Care
Drug: Lanadelumab — Lanadelumab administered as an intravenous (IV) infusion.
  Other Names: TAKHZYRO™; TAK-743
  Arms: Lanadelumab + Standard of Care
Drug: Lanadelumab placebo — Matching lanadelumab placebo (normal saline) administered as an intravenous (IV) infusion.
  Arms: Lanadelumab Placebo + Standard of Care
Drug: Zilucoplan — Zilucoplan administered as a subcutaneous (sc) injection in the abdomen, thigh, or upper arm.
  Arms: Zilucoplan + Standard of Care
Drug: Zilucoplan placebo — Matching zilucoplan placebo administered as a subcutaneous (sc) injection in the abdomen, thigh, or upper arm.
  Arms: Zilucoplan Placebo + Standard of Care

SUMMARY:
The primary objective of this study is to evaluate the time to confirmed clinical recovery in participants hospitalized with COVID-19. Candidate agents will be evaluated frequently for efficacy and safety, with candidate agents being added to and/or removed from the study on an ongoing basis, depending on the results of their evaluation.

DETAILED DESCRIPTION:
This adaptive, randomized, placebo-controlled platform study is designed to rapidly assess multiple candidate agents as treatments for COVID-19 in hospitalized patients. Candidate agents will be evaluated frequently (through ongoing monitoring) for futility and safety, with candidate agents being added to and/or removed from the study on an ongoing basis, depending on the results of their evaluation.

For inclusion, participants will need to be hospitalized with a clinical status of Grade 2 to Grade 5, as defined by the following Clinical Severity Status 8-Point Ordinal Scale:

1. Death
2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
3. Hospitalized, on noninvasive ventilation or high-flow oxygen devices
4. Hospitalized, requiring supplemental oxygen
5. Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care (COVID-19 related or otherwise)
6. Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care
7. Not hospitalized, limitation on activities and/or requiring home oxygen
8. Not hospitalized, no limitations on activities

Participants will be randomized equally to either the candidate agent plus standard of care (SoC) or placebo plus SoC in a double-blind fashion. Participants who are randomized to placebo plus SoC will subsequently be randomized equally to a matching placebo corresponding to an available agent whose sub-protocol the patient qualified for (ie, a 2-stage randomization). Each participant in the placebo plus SoC group will only receive one type of placebo. Randomization will be stratified by baseline clinical severity of 2 on the 8-point ordinal scale (yes/no) and remdesivir use at baseline (yes/no).

The study will evaluate each candidate agent separately as an add-on to the SoC to assess safety and efficacy. The comparator group for a candidate agent will include participants randomized to the placebo arm of any sub-protocol according to the following conditions:

* Apremilast sub-protocol: participants who were enrolled concurrently to apremilast and who would have been eligible for the apremilast sub-protocol.
* Lanadelumab sub-protocol: at a site where at least one participant was randomized to either lanadelumab active or placebo arms.
* Zilucoplan sub-protocol: at a site where at least one participant was randomized to either the zilucoplan active or placebo arms.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years of age) with active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection confirmed by laboratory tests and/or point of care tests (eg, commercial or public health assay, which is approved for emergency use). If no diagnostic test results are available that have been obtained during the previous 72 hours, then a test should be performed as part of the screening assessment.
* A score of Grade 2 (hospitalized, on invasive mechanical ventilation or ECMO), Grade 3 (hospitalized, on noninvasive ventilation or high-flow oxygen devices), Grade 4 (hospitalized, requiring supplemental oxygen), or Grade 5 (hospitalized, not requiring supplemental oxygen, requiring ongoing medical care [COVID-19 related or otherwise]), as defined by an 8 point ordinal scale.
* Male participants:

  * A male participant must agree to use contraception during the treatment period and for at least 6 weeks after the last dose of study treatment and refrain from donating sperm during this period.
* Female participants:

  * A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies:
  * Not a woman of childbearing potential (WOCBP). OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 6 weeks after the last dose of study treatment.
* Ability to provide informed consent signed by the study participant or legally authorized representative.
* Ability and willingness to participate in telephone/telemedicine follow-up visits if needed.
* Zilucoplan only: Antibiotic prophylaxis: all participants must be willing to take antibiotic prophylaxis concomitantly, starting with the first dose of zilucoplan or placebo.

Exclusion Criteria:

* Participant has any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the participant (eg, compromise their well-being) or that could prevent, limit, or confound the protocol-specified assessments (eg, participants unable to swallow study medication tablets).
* Stage 4 severe chronic kidney disease or requiring dialysis.
* Screening 12-lead electrocardiogram (ECG) with a measurable QTc interval according to Fridericia correction (QTcF) ≥ 500 ms.
* Anticipated transfer to another hospital that is not a study center within 72 hours.
* Participants who are currently pregnant or who are not willing to discontinue breastfeeding.
* Participants participating in another clinical study of an investigational medicinal product or other unapproved (or investigational) treatment for COVID-19.
* Active tuberculosis or a history of incompletely treated tuberculosis.
* Active, uncontrolled systemic bacterial or fungal infection(s).
* Apremilast only: Current treatment with apremilast, or another agent of similar mechanism of action, for any indication within 1 week prior to first dose of investigational product.
* Apremilast only: Concurrent use at screening or randomization of cytochrome P450 (CYP)3A inducers (eg, rifampin, phenobarbital, carbamazepine) within 1 week prior to first dose of investigational product.
* Apremilast only: Known hypersensitivity to apremilast or any excipients in formulation.
* Lanadelumab only: Known or suspected hypersensitivity to lanadelumab or any of its excipients.
* Lanadelumab only: Previous (within 3 months prior to baseline) or current use of immunomodulators (eg, methotrexate, azathioprine, 6-mercaptopurine, tumor necrosis factor [TNF] α inhibitor, Janus kinase [JAK] inhibitor, alpha-integrin inhibitor).
* Lanadelumab only: Known or suspected venous thromboembolism.
* Lanadelumab only: Previous (within 3 months [or 5 half-lives, whichever is greater] of screening) or current use of plasma kallikrein (pKal) inhibitor or bradykinin receptor blocker.
* Zilucoplan only: Participants with unresolved or suspected infection with Neisseria meningitidis or a past history of N. meningitidis (eg, in a complement-deficient patient).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (59):
- United States (21):
  - Pinnacle Research Group LLC, Anniston, Alabama
  - Good Samaritan Hospital, Bakersfield, California
  - Sharp Chula Vista Medical Center, Chula Vista, California
  - El Centro Regional Medical Center, El Centro, California
  - University of California Irvine Medical Center, Orange, California
  - Riverside Community Hospital, Riverside, California
  - University of California Davis Health System, Sacramento, California
  - National Institute of Clinical Research, South El Monte, California
  - UF Health Shands Hospital, Gainesville, Florida
  - Memorial Hospital Jacksonville, Jacksonville, Florida
  - Grady Health System, Atlanta, Georgia
  - Great Lakes Clinical Trials, Chicago, Illinois
  - The University of Iowa, Iowa City, Iowa
  - Harper University Hospital, Detroit, Michigan
  - Sinai Grace Hospital, Detroit, Michigan
  - Detroit Receiving Hospital, Royal Oak, Michigan
  - University of Tennessee Health Sciences Center, Memphis, Tennessee
  - Medical City Ft. Worth, Fort Worth, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Texoma Medical Center, Sherman, Texas
  - MultiCare Health System Institute for Research and Innovation, Tacoma, Washington
- Argentina (5):
  - Hospital San Juan de Dios, Ramos Mejía, Buenos Aires
  - Hospital General de Agudos Dr. J. M. Ramos Mejia, Ciudad Autonoma Buenos Aires
  - Hospital General de Agudos Dr. Ignacio Pirovano, Ciudad Autonoma Buenos Aires
  - Clinica Adventista Belgrano, Ciudad Autonoma Buenos Aires
  - Hospital Italiano de Rosario, Rosario
- Brazil (6):
  - Chronos Pesquisa Clinica, Brasília, Federal District
  - HC-UFG - Hospital das Clínicas da Universidade Federal de Goiás, Goiânia, Goiás
  - Santa Casa de Misericórdia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu, São Paulo
  - Praxis Pesquisa Médica, Santo André, São Paulo
- Hospital Base Osorno, Osorno, Chile
- Mexico (4):
  - Hospital General de Tijuana, Tijuana, Baja California Norte
  - Hospital Civil de Guadalajara Dr. Juan I. Menchaca, Guadalajara, Jalisco
  - Universidad Autonoma de Nuevo Leon, Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Hospital Civil de Culiacan, Culiacán, Sinaloa
- Russia (7):
  - TSBIH "Krasnoyarsk Interdistrict Clinical Hospital of Emergency Medical Care n.a. N.S. Karpovich, Krasnoyarsk
  - SBIH of Moscow "Infectious Clinical Hospital # 1 of Department of Healthcare of Moscow", Moscow
  - SPb SBIH "Alexandrovskaya City Hospital", Saint Petersburg
  - St-George Hospital, Saint Petersburg
  - SPb SBIH "Nikolaevskaya Hospital", Saint Petersburg
  - SPb SBIH "City Pokrovskaya Hospital", Saint Petersburg
  - SPb SBIH "City Hospital # 40 of Kurortnyi region", Sestroretsk
- South Africa (9):
  - Nelson Mandela Academic Clinical Research Unit (NeMACRU), Mthatha, Eastern Cape
  - Johese Clinical Research: Unitas, Centurion, Gauteng
  - MERC SiReN, Johannesburg, Gauteng
  - Drs Sarvan and Moodley, Durban, KwaZulu-Natal
  - Tread Research, Cape Town, Western Cape
  - Tiervlei Trial Centre, Cape Town, Western Cape
  - 2 Military Hospital Internal Medicine, Cape Town, Western Cape
  - Dr JM Engelbrecht Trial Site, Somerset West, Western Cape
  - Clinical Projects Research SA (PTY) LTD, Worcester, Western Cape
- Ukraine (6):
  - Communal Noncommercial Profit "Clinical City Hospital 16 of Dnipro Regional Council", Dnipro
  - CNE of Kharkov RC Reg Cl Infectious Hospital, Kharkiv
  - Communal Non-Commercial Medical Enterprise "O.T.Bohayevskyi Kremenchuk City Hospital #1", Kremenchuk
  - City Clinical infectious Hospital, Odesa
  - Municipal Non-Profit Enterprise Central City Hospital Of Rivne City Council, Rivne
  - CCH #1 Vinnytsia M.I.Pyrogov NMU Ch of Infectious Diseases, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This adaptive platform study consisted of 3 sub-protocols, each designed to assess a candidate agent as treatment for coronavirus disease 2019 (COVID-19) in hospitalized adult patients who had severe infection with acute respiratory syndrome coronavirus 2 (SARS-CoV-2), the virus that causes COVID-19.
  The control group for a candidate agent includes participants randomized to any matching placebo for a candidate agent if certain criteria were met (shared placebo).
Pre-assignment Details: Participants were initially randomized to an active candidate agent or generically to placebo plus standard of care (SoC) for sub-protocols for which they met eligibility. Participants randomized to placebo plus SoC were subsequently randomized equally to a matching placebo for an available candidate agent whose sub-protocol the participant qualified for. Randomization was stratified by baseline clinical severity of 2 on the 8-point ordinal scale (yes/no) and remdesivir use at baseline (yes/no).
Groups:
- Lanadelumab + Standard of Care: Participants randomized to receive lanadelumab 300 mg by intravenous infusion on Day 1, and a second dose administered on Day 4, in addition to standard of care.
- Lanadelumab Placebo + Standard of Care: Participants randomized to receive placebo to lanadelumab by intravenous infusion on Day 1, and a second dose administered on Day 4 in, addition to standard of care.
- Apremilast + Standard of Care: Participants randomized to received 30 mg apremilast orally twice a day (BID) in addition to standard of care treatment for 14 days or until hospital discharge, whichever occurred first.
- Apremilast Placebo + Standard of Care: Participants randomized to receive matching placebo to apremilast orally twice a day in addition to standard of care treatment for 14 days or until hospital discharge, whichever occurred first.
- Zilucoplan + Standard of Care: Participants randomized to receive 32.4 mg zilucoplan by subcutaneous injection every day for 14 days, or until discharge if discharge was before 14 days of treatment, in addition to standard of care.
- Zilucoplan Placebo + Standard of Care: Participants randomized to receive placebo to zilucoplan by subcutaneous injection every day for 14 days, or until discharge if discharge was before 14 days of treatment, in addition to standard of care.
Period: Overall Study
Arm/Group | Lanadelumab + Standard of Care | Lanadelumab Placebo + Standard of Care | Apremilast + Standard of Care | Apremilast Placebo + Standard of Care | Zilucoplan + Standard of Care | Zilucoplan Placebo + Standard of Care
Started | 28 | 1 | 194 | 184 | 100 | 8
Received Study Drug | 27 | 1 | 189 | 182 | 95 | 7
Full Analysis Set (For each sub-protocol the full analysis set includes all participants randomized to the sub-protocol candidate agent as well as all participants who were randomized to any placebo arm included in the control arm of the candidate agent (i.e. shared placebo). The control arm for analysis of a candidate agent includes participants enrolled in any placebo group, regardless of sub-protocol, if certain criteria were met.) | 28 | 34 (Includes participants randomized to this arm (1) and 32 participants from Apremilast Placebo + SOC group and 1 participant from Zilucoplan Placebo + SOC group.) | 194 | 190 (Includes participants randomized to this arm (184) and 1 participant from Lanadelumab Placebo + SOC group and 5 participants from Zilucoplan Placebo + SOC group.) | 100 | 75 (Includes participants randomized to this arm (8) and 1 participant from Lanadelumab Placebo + SOC group and 66 participants from the Apremilast Placebo + SOC group.)
Completed | 15 | 0 | 139 | 138 | 70 | 4
Not Completed | 13 | 1 | 55 | 46 | 30 | 4
Not completed — Death | 7 | 1 | 37 | 34 | 19 | 3
Not completed — Lost to Follow-up | 3 | 0 | 11 | 11 | 6 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 0 | 3 | 0
Not completed — Other | 3 | 0 | 1 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for the full analysis set, which includes all participants who were randomized to the sub-protocol candidate agent arm as well as all participants who were randomized to any placebo arm included in the control arm of the candidate agent. The Total number of participants (621) includes participants randomized to placebo and included in more than one placebo control group (106 participants); 515 unique participants were enrolled in the study.
Groups:
- Lanadelumab Placebo Control: Includes participants randomized to receive matching placebo to lanadelumab plus standard of care treatment as well as participants who were randomized to receive placebo to apremilast or placebo to zilucoplan plus standard of care treatment at a site that enrolled at least one participant in the lanadelumab sub-protocol.
- Apremilast + Standard of Care: Participants randomized to receive 30 mg apremilast orally twice a day (BID) in addition to standard of care treatment for 14 days or until hospital discharge, whichever occurred first.
- Apremilast Placebo Control: Includes participants randomized to receive matching placebo to apremilast plus standard of care treatment as well as participants who were randomized to receive placebo to lanadelumab or placebo to zilucoplan plus standard of care treatment at a site concurrently enrolling apremilast sub-protocol participants and who would have been eligible for the apremilast sub-protocol.
- Zilucoplan Placebo +Control: Includes participants randomized to receive matching placebo to zilucoplan plus standard of care treatment as well as participants who were randomized to receive placebo to lanadelumab or placebo to apremilast plus standard of care treatment at a site that enrolled at least one participant in the zilucoplan sub-protocol.
- Total: Total of all reporting groups
Arm/Group | Lanadelumab + Standard of Care | Lanadelumab Placebo Control | Apremilast + Standard of Care | Apremilast Placebo Control | Zilucoplan + Standard of Care | Zilucoplan Placebo +Control | Total
Number analyzed (Participants) | 28 | 34 | 194 | 190 | 100 | 75 | 621
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data are reported separately for each subprotocol so as not to double-count participants in the shared placebo control groups.
  years
    Lanadelumab Sub-protocol: number analyzed (Participants) | 28 | 34 | 0 | 0 | 0 | 0 | 62
    Lanadelumab Sub-protocol | 53.4 (15.34) | 59.6 (13.50) |  |  |  |  | 56.8 (14.57)
    Apremilast Sub-protocol: number analyzed (Participants) | 0 | 0 | 194 | 190 | 0 | 0 | 384
    Apremilast Sub-protocol |  |  | 57.2 (13.84) | 55.7 (13.37) |  |  | 56.5 (13.61)
    Zilucoplan Sub-protocol: number analyzed (Participants) | 0 | 0 | 0 | 0 | 100 | 75 | 175
    Zilucoplan Sub-protocol |  |  |  |  | 53.2 (14.13) | 58.4 (13.62) | 55.4 (14.11)
Age, Customized [Count of Participants; unit: Participants] — Population: Age data are reported separately for each subprotocol so as not to double-count participants in the shared placebo control groups.
  Participants
    Lanadelumab Sub-protocol: number analyzed (Participants) | 28 | 34 | 0 | 0 | 0 | 0 | 62
    Lanadelumab Sub-protocol: ≥ 18 to ≤ 49 years | 13 | 8 |  |  |  |  | 21
    Lanadelumab Sub-protocol: ≥ 50 to ≤ 64 years | 7 | 15 |  |  |  |  | 22
    Lanadelumab Sub-protocol: ≥ 65 to ≤ 84 years | 8 | 10 |  |  |  |  | 18
    Lanadelumab Sub-protocol: ≥ 85 years | 0 | 1 |  |  |  |  | 1
    Apremilast Sub-protocol: number analyzed (Participants) | 0 | 0 | 194 | 190 | 0 | 0 | 384
    Apremilast Sub-protocol: ≥ 18 to ≤ 49 years |  |  | 51 | 56 |  |  | 107
    Apremilast Sub-protocol: ≥ 50 to ≤ 64 years |  |  | 76 | 81 |  |  | 157
    Apremilast Sub-protocol: ≥ 65 to ≤ 84 years |  |  | 64 | 52 |  |  | 116
    Apremilast Sub-protocol: ≥ 85 years |  |  | 3 | 1 |  |  | 4
    Zilucoplan Sub-protocol: number analyzed (Participants) | 0 | 0 | 0 | 0 | 100 | 75 | 175
    Zilucoplan Sub-protocol: ≥ 18 to ≤ 49 years |  |  |  |  | 45 | 19 | 64
    Zilucoplan Sub-protocol: ≥ 50 to ≤ 64 years |  |  |  |  | 36 | 29 | 65
    Zilucoplan Sub-protocol: ≥ 65 to ≤ 84 years |  |  |  |  | 16 | 26 | 42
    Zilucoplan Sub-protocol: ≥ 85 years |  |  |  |  | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex data are reported separately for each subprotocol so as not to double-count participants in the shared placebo control groups.
  Participants
    Lanadelumab Sub-protocol: number analyzed (Participants) | 28 | 34 | 0 | 0 | 0 | 0 | 62
    Lanadelumab Sub-protocol: Female | 11 | 9 | 0 | 0 | 0 | 0 | 20
    Lanadelumab Sub-protocol: Male | 17 | 25 | 0 | 0 | 0 | 0 | 42
    Apremilast Sub-protocol: number analyzed (Participants) | 0 | 0 | 194 | 190 | 0 | 0 | 384
    Apremilast Sub-protocol: Female | 0 | 0 | 84 | 72 | 0 | 0 | 156
    Apremilast Sub-protocol: Male | 0 | 0 | 110 | 118 | 0 | 0 | 228
    Zilucoplan Sub-protocol: number analyzed (Participants) | 0 | 0 | 0 | 0 | 100 | 75 | 175
    Zilucoplan Sub-protocol: Female | 0 | 0 | 0 | 0 | 34 | 28 | 62
    Zilucoplan Sub-protocol: Male | 0 | 0 | 0 | 0 | 66 | 47 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data are reported separately for each subprotocol so as not to double-count participants in the shared placebo control groups.
  Participants
    Lanadelumab Sub-protocol: number analyzed (Participants) | 28 | 34 | 0 | 0 | 0 | 0 | 62
    Lanadelumab Sub-protocol: Hispanic or Latino | 18 | 19 |  |  |  |  | 37
    Lanadelumab Sub-protocol: Not Hispanic or Latino | 10 | 15 |  |  |  |  | 25
    Lanadelumab Sub-protocol: Unknown or Not Reported | 0 | 0 |  |  |  |  | 0
    Apremilast Sub-protocol: number analyzed (Participants) | 0 | 0 | 194 | 190 | 0 | 0 | 384
    Apremilast Sub-protocol: Hispanic or Latino |  |  | 75 | 72 |  |  | 147
    Apremilast Sub-protocol: Not Hispanic or Latino |  |  | 108 | 112 |  |  | 220
    Apremilast Sub-protocol: Unknown or Not Reported |  |  | 11 | 6 |  |  | 17
    Zilucoplan Sub-protocol: number analyzed (Participants) | 0 | 0 | 0 | 0 | 100 | 75 | 175
    Zilucoplan Sub-protocol: Hispanic or Latino |  |  |  |  | 65 | 32 | 97
    Zilucoplan Sub-protocol: Not Hispanic or Latino |  |  |  |  | 35 | 43 | 78
    Zilucoplan Sub-protocol: Unknown or Not Reported |  |  |  |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race data are reported separately for each subprotocol so as not to double-count participants in the shared placebo control groups.
  Participants
    Lanadelumab Sub-protocol: number analyzed (Participants) | 28 | 34 | 0 | 0 | 100 | 75 | 237
    Lanadelumab Sub-protocol: American Indian or Alaska Native | 1 | 0 |  |  | 3 | 1 | 5
    Lanadelumab Sub-protocol: Asian | 0 | 0 |  |  | 3 | 5 | 8
    Lanadelumab Sub-protocol: Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0 | 0 | 0
    Lanadelumab Sub-protocol: Black or African American | 3 | 2 |  |  | 5 | 5 | 15
    Lanadelumab Sub-protocol: White | 20 | 28 |  |  | 75 | 58 | 181
    Lanadelumab Sub-protocol: More than one race | 2 | 1 |  |  | 8 | 2 | 13
    Lanadelumab Sub-protocol: Unknown or Not Reported | 2 | 3 |  |  | 6 | 4 | 15
    Apremilast Sub-protocol: number analyzed (Participants) | 0 | 0 | 194 | 190 | 0 | 0 | 384
    Apremilast Sub-protocol: American Indian or Alaska Native |  |  | 0 | 1 |  |  | 1
    Apremilast Sub-protocol: Asian |  |  | 11 | 7 |  |  | 18
    Apremilast Sub-protocol: Native Hawaiian or Other Pacific Islander |  |  | 0 | 1 |  |  | 1
    Apremilast Sub-protocol: Black or African American |  |  | 9 | 9 |  |  | 18
    Apremilast Sub-protocol: White |  |  | 151 | 151 |  |  | 302
    Apremilast Sub-protocol: More than one race |  |  | 4 | 7 |  |  | 11
    Apremilast Sub-protocol: Unknown or Not Reported |  |  | 19 | 14 |  |  | 33
    Zilucoplan Sub-protocol: number analyzed (Participants) | 0 | 0 | 0 | 0 | 100 | 75 | 175
    Zilucoplan Sub-protocol: American Indian or Alaska Native |  |  |  |  | 3 | 1 | 4
    Zilucoplan Sub-protocol: Asian |  |  |  |  | 3 | 5 | 8
    Zilucoplan Sub-protocol: Native Hawaiian or Other Pacific Islander |  |  |  |  | 0 | 0 | 0
    Zilucoplan Sub-protocol: Black or African American |  |  |  |  | 5 | 5 | 10
    Zilucoplan Sub-protocol: White |  |  |  |  | 75 | 58 | 133
    Zilucoplan Sub-protocol: More than one race |  |  |  |  | 8 | 2 | 10
    Zilucoplan Sub-protocol: Unknown or Not Reported |  |  |  |  | 6 | 4 | 10
Region [Count of Participants; unit: Participants] — Geographic regions are: North America (USA), Latin America (Argentina, Brazil, Chile, and Mexico), Eastern Europe (Russian Federation and Ukraine), and Rest of the World (South Africa). Population: Region data are reported separately for each subprotocol so as not to double-count participants in the shared placebo control groups.
  Participants
    Lanadelumab Sub-protocol: number analyzed (Participants) | 28 | 34 | 0 | 0 | 0 | 0 | 62
    Lanadelumab Sub-protocol: North America | 9 | 9 |  |  |  |  | 18
    Lanadelumab Sub-protocol: Latin America | 18 | 20 |  |  |  |  | 38
    Lanadelumab Sub-protocol: Eastern Europe | 0 | 0 |  |  |  |  | 0
    Lanadelumab Sub-protocol: Rest of the World | 1 | 5 |  |  |  |  | 6
    Apremilast Sub-protocol: number analyzed (Participants) | 0 | 0 | 194 | 190 | 0 | 0 | 384
    Apremilast Sub-protocol: North America |  |  | 53 | 60 |  |  | 113
    Apremilast Sub-protocol: Latin America |  |  | 60 | 50 |  |  | 110
    Apremilast Sub-protocol: Eastern Europe |  |  | 51 | 53 |  |  | 104
    Apremilast Sub-protocol: Rest of the World |  |  | 30 | 27 |  |  | 57
    Zilucoplan Sub-protocol: number analyzed (Participants) | 0 | 0 | 0 | 0 | 100 | 75 | 175
    Zilucoplan Sub-protocol: North America |  |  |  |  | 26 | 10 | 36
    Zilucoplan Sub-protocol: Latin America |  |  |  |  | 65 | 33 | 98
    Zilucoplan Sub-protocol: Eastern Europe |  |  |  |  | 6 | 14 | 20
    Zilucoplan Sub-protocol: Rest of the World |  |  |  |  | 3 | 18 | 21
Remdesivir Use at Baseline [Count of Participants; unit: Participants] — Randomization was stratified by remdesivir use at baseline (yes or no), based on data captured on the interactive web response system (IWRS). Population: Data are reported separately for each subprotocol so as not to double-count participants in the shared placebo control groups.
  Participants
    Lanadelumab Sub-protocol: number analyzed (Participants) | 28 | 34 | 0 | 0 | 0 | 0 | 62
    Lanadelumab Sub-protocol: Yes | 7 | 5 |  |  |  |  | 12
    Lanadelumab Sub-protocol: No | 21 | 29 |  |  |  |  | 50
    Apremilast Sub-protocol: number analyzed (Participants) | 0 | 0 | 194 | 190 | 0 | 0 | 384
    Apremilast Sub-protocol: Yes |  |  | 45 | 44 |  |  | 89
    Apremilast Sub-protocol: No |  |  | 149 | 146 |  |  | 295
    Zilucoplan Sub-protocol: number analyzed (Participants) | 0 | 0 | 0 | 0 | 100 | 75 | 175
    Zilucoplan Sub-protocol: Yes |  |  |  |  | 22 | 9 | 31
    Zilucoplan Sub-protocol: No |  |  |  |  | 78 | 66 | 144
Clinical Severity Score of 2 [Count of Participants; unit: Participants] — Randomization was stratified by ordinal scale clinical severity score of Grade 2 vs Grade 3-5 per IWRS:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or ECMO
  3. Hospitalized, on noninvasive ventilation or high-flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care
  6. Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities Population: Data are reported separately for each subprotocol so as not to double-count participants in the shared placebo control groups.
  Participants
    Lanadelumab Sub-protocol: number analyzed (Participants) | 28 | 34 | 0 | 0 | 0 | 0 | 62
    Lanadelumab Sub-protocol: Yes (Grade 2) | 3 | 4 |  |  |  |  | 7
    Lanadelumab Sub-protocol: No (Grade 3-5) | 25 | 30 |  |  |  |  | 55
    Apremilast Sub-protocol: number analyzed (Participants) | 0 | 0 | 194 | 190 | 0 | 0 | 384
    Apremilast Sub-protocol: Yes (Grade 2) |  |  | 11 | 9 |  |  | 20
    Apremilast Sub-protocol: No (Grade 3-5) |  |  | 183 | 181 |  |  | 364
    Zilucoplan Sub-protocol: number analyzed (Participants) | 0 | 0 | 0 | 0 | 100 | 75 | 175
    Zilucoplan Sub-protocol: Yes (Grade 2) |  |  |  |  | 8 | 6 | 14
    Zilucoplan Sub-protocol: No (Grade 3-5) |  |  |  |  | 92 | 69 | 161

OUTCOME MEASURES:

1. Primary Outcome: Lanadelumab Sub-protocol: Time to Confirmed Clinical Recovery Without Rehospitalization Through Day 29
Description: Confirmed clinical recovery means the participant is fit for discharge from hospital, defined by achieving a score of 6 (hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care), 7 (not hospitalized, limitation on activities and/or requiring home oxygen), or 8 (not hospitalized, no limitations on activities) on the clinical severity status 8-point ordinal scale, without being re-hospitalized prior to Day 29.
  The Kaplan-Meier estimate of the time to confirmed clinical recovery through Day 29, without re-hospitalization through Day 29, was calculated from Study Day 1 to the earliest date on which the participant had a score of 6, 7, or 8 up to Day 29. Participants who never reached a score of 6, 7, or 8 on the clinical severity status 8-point ordinal scale before or on Day 29 were censored at Day 29. Participants who discontinued from the study before or on Day 29 were censored at time of discontinuation from study.
Time Frame: Day 1 (the day of the first dose of study drug for randomized participants who received at least one dose of study drug or the day of randomization for randomized participants who did not receive any study drug) to Day 29
Population: The lanadelumab sub-protocol primary analysis set includes all participants who were randomized to lanadelumab as well as all participants who were randomized to any placebo arm included in the control arm for lanadelumab with a baseline clinical severity status of Grade 3 to Grade 5 on the clinical severity status 8-point ordinal scale.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Lanadelumab + Standard of Care | Lanadelumab Placebo Control
Number analyzed (Participants) | 25 | 30
days | 10.0 [5.00 to NA] — Not estimable due to the low number of events | 15.5 [8.00 to NA] — Not estimable due to the low number of events
Statistical Analysis 1: Comparison: Lanadelumab + Standard of Care vs Lanadelumab Placebo Control; Test type: Superiority; p = 0.6672, Stratified log-rank test; Stratified by baseline score of 2 on the ordinal scale for clinical severity (yes/no), remdesivir use at baseline (yes/no), and geographic region; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.59 to 2.35] — Hazard ratio (Lanadelumab vs. placebo) from a Cox regression model including baseline clinical severity of 2 on the ordinal scale for clinical severity (yes/no), remdesivir use at baseline (yes/no), geographic region, and treatment arm as factors

2. Primary Outcome: Apremilast Sub-protocol: Time to Confirmed Clinical Recovery Without Rehospitalization Through Day 29
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The apremilast full analysis set (FAS) includes all participants who were randomized to the apremilast arm as well as all participants who were randomized to any placebo arm included in the control arm for apremilast.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Apremilast + Standard of Care | Apremilast Placebo Control
Number analyzed (Participants) | 194 | 190
days | 14.0 [11.00 to 15.00] | 14.0 [11.00 to 15.00]
Statistical Analysis 1: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Test type: Superiority; p = 0.8779, Stratified log-rank test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.77 to 1.24] — Hazard ratio (apremilast vs. placebo) from a Cox regression model including baseline clinical severity of 2 on the ordinal scale for clinical severity (yes/no), remdesivir use at baseline (yes/no), geographic region, and treatment arm as factors

3. Primary Outcome: Zilucoplan Sub-protocol: Time to Confirmed Clinical Recovery Without Rehospitalization Through Day 29
Description: as for outcome 1
Time Frame: as for outcome 1
Population: The zilucoplan full analysis set includes all participants who were randomized to the zilucoplan arm as well as all participants who were randomized to any placebo arm included in the control arm for zilucoplan.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Zilucoplan Placebo Control: Includes participants randomized to receive matching placebo to zilucoplan plus standard of care treatment as well as participants who were randomized to receive placebo to lanadelumab or placebo to apremilast plus standard of care treatment at a site that enrolled at least one participant in the zilucoplan sub-protocol.
Arm/Group | Zilucoplan + Standard of Care | Zilucoplan Placebo Control
Number analyzed (Participants) | 100 | 75
days | 14.0 [11.00 to 22.0] | 15.0 [11.00 to 22.00]

4. Secondary Outcome: Lanadelumab Sub-protocol: Percentage of Participants Who Achieved Oxygen-Free Recovery at Day 29
Description: Oxygen-free recovery at Day 29 is defined as being alive, discharged, and not receiving supplemental oxygen at Day 29. Participants who reached a score of 7 on the ordinal scale for clinical severity who were discharged to hospice care before or on Day 29 were considered as not discharged at Day 29. Participants with a missing oxygen-free recovery status at Day 29 were considered as not having an oxygen-free recovery.
Time Frame: Day 29
Population: Lanadelumab sub-protocol primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanadelumab + Standard of Care | Lanadelumab Placebo Control
Number analyzed (Participants) | 25 | 30
percentage of participants | 52.0 [31.31 to 72.20] | 56.7 [37.43 to 74.54]

5. Secondary Outcome: Lanadelumab Sub-protocol: Percentage of Participants With a ≥ 2-point Improvement From Baseline or Fit for Discharge on the Clinical Severity Status 8-Point Ordinal Scale at Day 29
Description: Fit for discharge is defined as achieving a score of 6, 7, or 8 on the clinical severity status 8-point ordinal scale. Participants with an ordinal scale score of 7 must not have been discharged to hospice care to be considered as fit for discharge. Participants with a missing clinical severity score at Day 29 were considered as not having met the event at Day 29.
  The clinical severity status 8-point ordinal scale scores are:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. Hospitalized, on noninvasive ventilation or high-flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities
Time Frame: Baseline (Day 1) and Day 29
Population: Lanadelumab sub-protocol primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanadelumab + Standard of Care | Lanadelumab Placebo Control
Number analyzed (Participants) | 25 | 30
percentage of participants | 72.0 [50.61 to 87.93] | 63.3 [43.86 to 80.07]

6. Secondary Outcome: Lanadelumab Sub-protocol: Percentage of Participants Who Died Before or on Day 29
Description: All-cause mortality is death due to any cause. Participants with an unknown alive/death status on Day 29 were considered alive for this analysis, with the exception of patients with a score of 7 who were discharged to hospice care before or on Day 29.
Time Frame: Day 1 to Day 29
Population: Lanadelumab sub-protocol primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanadelumab + Standard of Care | Lanadelumab Placebo Control
Number analyzed (Participants) | 25 | 30
percentage of participants | 32.0 [14.95 to 53.50] | 30.0 [14.73 to 49.40]

7. Secondary Outcome: Lanadelumab Sub-protocol: Clinical Severity Status 8-Point Ordinal Scale Score at Days 8, 15, and 29
Description: The clinical severity status 8-point ordinal scale scores are:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. Hospitalized, on noninvasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities
  Participants with a score of 7 who were discharged to hospice care are counted with participants with a score of 1 (death) for this endpoint.
Time Frame: Day 8, Day 15, and Day 29
Population: Lanadelumab sub-protocol primary analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab + Standard of Care | Lanadelumab Placebo Control
Number analyzed (Participants) | 25 | 30
Participants
  Day 8: 1 (Death or discharged to hospice care) | 3 | 3
  Day 8: 2 (Hospitalized on invasive mechanical ventilation or ECMO) | 4 | 6
  Day 8: 3 (Hospitalized on noninvasive ventilation or high-flow oxygen devices) | 3 | 4
  Day 8: 4 (Hospitalized, requiring supplemental oxygen) | 2 | 6
  Day 8: 5 (Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care) | 1 | 0
  Day 8: 6 (Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care) | 1 | 1
  Day 8: 7 (Not hospitalized, limitation on activities and/or requiring home oxygen) | 2 | 3
  Day 8: 8 (Not hospitalized, no limitations on activities) | 8 | 7
  Day 8: Missing | 1 | 0
  Day 15: 1 (Death or discharged to hospice care) | 3 | 7
  Day 15: 2 (Hospitalized on invasive mechanical ventilation or ECMO) | 3 | 4
  Day 15: 3 (Hospitalized on noninvasive ventilation or high-flow oxygen devices) | 1 | 0
  Day 15: 4 (Hospitalized, requiring supplemental oxygen) | 0 | 2
  Day 15: 5 (Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care) | 0 | 0
  Day 15: 6 (Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care) | 0 | 1
  Day 15: 7 (Not hospitalized, limitation on activities and/or requiring home oxygen) | 5 | 3
  Day 15: 8 (Not hospitalized, no limitations on activities) | 12 | 13
  Day 15: Missing | 1 | 0
  Day 29: 1 (Death or discharged to hospice care) | 7 | 9
  Day 29: 2 (Hospitalized on invasive mechanical ventilation or ECMO) | 0 | 2
  Day 29: 3 (Hospitalized on noninvasive ventilation or high-flow oxygen devices) | 0 | 0
  Day 29: 4 (Hospitalized, requiring supplemental oxygen) | 0 | 0
  Day 29: 5 (Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care) | 0 | 0
  Day 29: 6 (Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care) | 0 | 0
  Day 29: 7 (Not hospitalized, limitation on activities and/or requiring home oxygen) | 5 | 6
  Day 29: 8 (Not hospitalized, no limitations on activities) | 12 | 13
  Day 29: Missing | 1 | 0

8. Secondary Outcome: Lanadelumab Sub-protocol: Worst Post-Baseline Score on Clinical Severity Status 8-point Ordinal Scale From Baseline to Day 29
Description: The worst post-baseline score (lower scores are worse) through Day 29 in the clinical severity status 8-point ordinal scale, derived from all scores recorded after baseline up to and including Day 29. Participants with a score of 7 discharged to hospice care are considered as having a score of 1 (death) instead of a score of 7 for this endpoint.
  The clinical severity status 8-point ordinal scale scores are:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or ECMO
  3. Hospitalized, on noninvasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities
Time Frame: Day 2 to Day 29
Population: Lanadelumab sub-protocol primary analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab + Standard of Care | Lanadelumab Placebo Control
Number analyzed (Participants) | 25 | 30
Participants
  1 (Death or discharged to hospice care) | 8 | 9
  2 (Hospitalized on invasive mechanical ventilation or ECMO) | 0 | 4
  3 (Hospitalized on noninvasive ventilation or high-flow oxygen devices) | 6 | 5
  4 (Hospitalized, requiring supplemental oxygen) | 8 | 11
  5 (Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care) | 1 | 0
  6 (Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care) | 0 | 0
  7 (Not hospitalized, limitation on activities and/or requiring home oxygen) | 0 | 0
  8 (Not hospitalized, no limitations on activities) | 1 | 1
  Missing | 1 | 0

9. Secondary Outcome: Lanadelumab Sub-protocol: Number of Intensive Care Unit (ICU) Days From Day 1 Through Day 29
Description: Number of ICU days is the sum of the duration of any episode of ICU admission between Day 1 and Day 29, both inclusive. The number of ICU days of participants who died before or on Day 29 as well as of participants with a score of 7 on the clinical severity status 8-point ordinal scale who were discharged to hospice care by Day 29 was set to 30 (worst possible outcome).
Time Frame: Day 1 to Day 29
Population: Lanadelumab sub-protocol primary analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab + Standard of Care | Lanadelumab Placebo Control
Number analyzed (Participants) | 25 | 30
Participants
  0 days | 13 | 10
  1 day | 1 | 1
  3 days | 0 | 1
  5 days | 0 | 1
  6 days | 0 | 2
  8 days | 1 | 3
  11 days | 2 | 0
  13 days | 1 | 1
  15 days | 0 | 1
  21 days | 0 | 1
  30 days (death or discharged to hospice care) | 7 | 9

10. Secondary Outcome: Lanadelumab Sub-protocol: Number of Invasive Mechanical Ventilator Days From Day 1 Through Day 29
Description: Number of invasive mechanical ventilator days is the sum of the duration of any episode of invasive mechanical ventilator admission between Day 1 and Day 29, both inclusive. The number of invasive mechanical ventilator days of participants who died before or on Day 29 as well as of participants with a score of 7 on the clinical severity status 8-point ordinal scale who were discharged to hospice care by Day 29 was set to 30.
Time Frame: Day 1 to Day 29
Population: Lanadelumab sub-protocol primary analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab + Standard of Care | Lanadelumab Placebo Control
Number analyzed (Participants) | 25 | 30
Participants
  0 days | 17 | 18
  6 days | 0 | 1
  16 days | 0 | 1
  24 days | 0 | 1
  30 days (death or discharged to hospice care) | 8 | 9

11. Secondary Outcome: Lanadelumab Sub-protocol: Percentage of Participants Who Achieved Clinical Recovery by Days 8, 15, and 29
Description: Clinical recovery is defined as being fit for discharge, i.e., the achievement of a score of 6, 7, or 8 on the clinical severity status 8-point ordinal scale. Participants with a score of 7 discharged to hospice care were not considered fit for discharge. Participants who discontinued the study on or before Days 8, 15, or 29 or with a missing clinical recovery status were considered as not having clinical recovery at each respective time point.
  Clinical severity status 8-point ordinal scale:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or ECMO
  3. Hospitalized, on noninvasive ventilation or high-flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care
  6. Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities
Time Frame: Day 8, Day 15, and Day 29
Population: Lanadelumab sub-protocol primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanadelumab + Standard of Care | Lanadelumab Placebo Control
Number analyzed (Participants) | 25 | 30
percentage of participants
  Day 8 | 44.0 [24.40 to 65.07] | 36.7 [19.93 to 56.14]
  Day 15 | 56.0 [34.93 to 75.60] | 56.7 [37.43 to 75.54]
  Day 29 | 60.0 [38.67 to 78.87] | 63.3 [43.86 to 80.07]

12. Secondary Outcome: Lanadelumab Sub-protocol: Percentage of Participants Who Achieved Sustained Clinical Recovery
Description: Sustained clinical recovery is defined as being fit for discharge (achieving a score of 6, 7, or 8 on the clinical severity status 8-point ordinal scale) by Day 29, without re-hospitalization by Day 60. Participants with a score of 7 discharged to hospice care were not considered fit for discharge. Participants who died or discontinued from study or with a missing clinical recovery status at Day 60 were not considered having sustained clinical recovery.
  Clinical severity status 8-point ordinal scale:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or ECMO
  3. Hospitalized, on noninvasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care
  6. Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities
Time Frame: Day 60
Population: Lanadelumab sub-protocol primary analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lanadelumab + Standard of Care | Lanadelumab Placebo Control
Number analyzed (Participants) | 25 | 30
percentage of participants | 40.0 [21.13 to 61.33] | 56.7 [37.43 to 74.54]

13. Secondary Outcome: Lanadelumab Sub-protocol: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to study treatment. A TEAE is an AE that occurs after the first dose of study drug. A Serious AE is any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of hospitalization, resulted in persistent disability/incapacity, a congenital anomaly/birth defect, or an important medical event that may jeopardize the patient or require intervention to prevent an outcome listed above.
  The Investigator assessed the intensity of each AE according to the Common Terminology Criteria for Adverse Events (CTCAE):
  * Grade 1 Mild; asymptomatic or mild symptoms;
  * Grade 2 Moderate; minimal, local or noninvasive intervention indicated;
  * Grade 3 Severe or medically significant, not immediately life-threatening;
  * Grade 4 Life-threatening; urgent intervention indicated;
  * Grade 5 Death due to AE.
Time Frame: From first dose of study drug to end of study (Day 60)
Population: Lanadelumab safety analysis set included all participants in the lanadelumab FAS who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Lanadelumab + Standard of Care: Participants received lanadelumab 300 mg by intravenous infusion on Day 1, and a second dose administered on Day 4, in addition to standard of care.
- Lanadelumab Placebo Control: Includes participants who received matching placebo to lanadelumab plus standard of care treatment as well as participants who received placebo to apremilast or placebo to zilucoplan plus standard of care treatment at a site that enrolled at least one participant in the lanadelumab sub-protocol.
- Lanadelumab Placebo + Standard of Care: Participants received placebo to lanadelumab by intravenous infusion on Day 1, and a second dose administered on Day 4 in, addition to standard of care.
Arm/Group | Lanadelumab + Standard of Care | Lanadelumab Placebo Control | Lanadelumab Placebo + Standard of Care
Number analyzed (Participants) | 27 | 34 | 1
Participants
  Any treatment-emergent adverse event (TEAE) | 17 | 22 | 1
  TEAE with a CTCAE grade ≥ 3 | 11 | 18 | 1
  Serious TEAE | 11 | 18 | 1
  TEAE leading to dose modification | 2 | 3 | 0
  TEAE leading to discontinuation of study drug | 1 | 5 | 0

14. Secondary Outcome: Apremilast Sub-protocol: Percentage of Participants Who Achieved Oxygen-Free Recovery at Day 29
Description: as for outcome 4
Time Frame: Day 29
Population: Apremilast sub-protocol full analysis set
Measure: Number; unit: percentage of participants
Groups:
- Apremilast + Standard of Care: Participants randomized to receive 30 mg apremilast orally twice a day in addition to standard of care treatment for 14 days or until hospital discharge, whichever occurred first.
Arm/Group | Apremilast + Standard of Care | Apremilast Placebo Control
Number analyzed (Participants) | 194 | 190
percentage of participants | 59.8 | 63.7
Statistical Analysis 1: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Test type: Other; p = 0.3773, Regression, Logistic; Risk Difference (RD) = -4.0, 95% CI 2-sided [-12.9 to 4.9] — Risk difference is from a logistic regression including the baseline clinical severity of 2 on the ordinal scale for clinical severity (yes/no), remdesivir use at baseline (yes/no), geographic region, and treatment arm as factors
Statistical Analysis 2: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Test type: Other; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.52 to 1.28] — Odds ratio (apremilast vs. placebo) is from a logistic regression including the baseline clinical severity of 2 on the ordinal scale for clinical severity (yes/no), remdesivir use at baseline (yes/no), geographic region, and treatment arm as factors

15. Secondary Outcome: Apremilast Sub-protocol: Percentage of Participants With a ≥ 2-point Improvement From Baseline or Fit for Discharge on the Clinical Severity Status 8-Point Ordinal Scale at Day 29
Description: Fit for discharge is defined as achieving a score of 6, 7, or 8 on the clinical severity status 8-point ordinal scale. Participants with an ordinal scale score of 7 must not have been discharged to hospice care to be considered as fit for discharge. Participants with a missing clinical severity score at Day 29 were considered as not having met the event at Day 29.
  The clinical severity status 8-point ordinal scale scores are:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or ECMO
  3. Hospitalized, on noninvasive ventilation or high-flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities
Time Frame: Baseline (Day 1) and Day 29
Population: Apremilast sub-protocol full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast + Standard of Care | Apremilast Placebo Control
Number analyzed (Participants) | 194 | 190
percentage of participants | 74.7 | 77.9
Statistical Analysis 1: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Test type: Other; p = 0.4846, Regression, Logistic; Risk Difference (RD) = -2.9, 95% CI 2-sided [-11.2 to 5.3] — Risk difference is from a logistic regression including baseline clinical severity of 2 on the ordinal scale for clinical severity (yes/no), remdesivir use at baseline (yes/no), geographic region, and treatment arm as factors
Statistical Analysis 2: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Test type: Other; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.51 to 1.37] — Odds ratio (apremilast vs. placebo) is from a logistic regression including baseline clinical severity of 2 on the ordinal scale for clinical severity (yes/no), remdesivir use at baseline (yes/no), geographic region, and treatment arm as factors

16. Secondary Outcome: Apremilast Sub-protocol: Percentage of Participants Who Died Before or on Day 29
Description: as for outcome 6
Time Frame: Day 1 to Day 29
Population: Apremilast sub-protocol full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast + Standard of Care | Apremilast Placebo Control
Number analyzed (Participants) | 194 | 190
percentage of participants | 17.5 | 17.4
Statistical Analysis 1: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Test type: Other; p = 0.9665, Regression, Logistic; Risk Difference (RD) = 0.2, 95% CI 2-sided [-7.3 to 7.6] — [estimate comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Test type: Other; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.59 to 1.74] — [estimate comment as in outcome 14, analysis 2]

17. Secondary Outcome: Apremilast Sub-protocol: Clinical Severity Status 8-Point Ordinal Scale Score at Days 8, 15, and 29
Description: as for outcome 7
Time Frame: Day 8, Day 15, and Day 29
Population: Apremilast sub-protocol full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast + Standard of Care | Apremilast Placebo Control
Number analyzed (Participants) | 194 | 190
Participants
  Day 8: 1 (Death or discharged to hospice care) | 11 | 8
  Day 8: 2 (Hospitalized on invasive mechanical ventilation or ECMO) | 22 | 20
  Day 8: 3 (Hospitalized on noninvasive ventilation or high-flow oxygen devices) | 25 | 26
  Day 8: 4 (Hospitalized, requiring supplemental oxygen) | 26 | 26
  Day 8: 5 (Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care) | 31 | 40
  Day 8: 6 (Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care) | 0 | 1
  Day 8: 7 (Not hospitalized, limitation on activities and/or requiring home oxygen) | 36 | 33
  Day 8: 8 (Not hospitalized, no limitations on activities) | 38 | 34
  Day 8: Missing | 5 | 2
  Day 15: 1 (Death or discharged to hospice care) | 22 | 24
  Day 15: 2 (Hospitalized on invasive mechanical ventilation or ECMO) | 16 | 13
  Day 15: 3 (Hospitalized on noninvasive ventilation or high-flow oxygen devices) | 9 | 9
  Day 15: 4 (Hospitalized, requiring supplemental oxygen) | 9 | 8
  Day 15: 5 (Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care) | 10 | 5
  Day 15: 6 (Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care) | 0 | 2
  Day 15: 7 (Not hospitalized, limitation on activities and/or requiring home oxygen) | 46 | 48
  Day 15: 8 (Not hospitalized, no limitations on activities) | 78 | 79
  Day 15: Missing | 4 | 2
  Day 29: 1 (Death or discharged to hospice care) | 34 | 31
  Day 29: 2 (Hospitalized on invasive mechanical ventilation or ECMO) | 6 | 6
  Day 29: 3 (Hospitalized on noninvasive ventilation or high-flow oxygen devices) | 0 | 3
  Day 29: 4 (Hospitalized, requiring supplemental oxygen) | 6 | 1
  Day 29: 5 (Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care) | 0 | 1
  Day 29: 6 (Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care) | 0 | 2
  Day 29: 7 (Not hospitalized, limitation on activities and/or requiring home oxygen) | 34 | 40
  Day 29: 8 (Not hospitalized, no limitations on activities) | 110 | 104
  Day 29: Missing | 4 | 2
Statistical Analysis 1: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Day 8; Test type: Other; p = 0.9119, Proportional odds model; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.71 to 1.46] — Odds ratio (Apremilast vs. Placebo) from a proportional odds model including the baseline clinical severity of 2 on the 8-point ordinal scale for clinical severity (yes/no), remdesivir use at baseline (yes/no), region, and treatment arm as factors
Statistical Analysis 2: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Day 15; Test type: Other; p = 0.6475, Proportional odds model; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.75 to 1.58] — [estimate comment as in outcome 17, analysis 1]
Statistical Analysis 3: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Day 29; Test type: Other; p = 0.9071, Proportional odds model; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.64 to 1.48] — [estimate comment as in outcome 17, analysis 1]

18. Secondary Outcome: Apremilast Sub-protocol: Worst Post-Baseline Score on Clinical Severity Status 8-Point Ordinal Scale From Baseline to Day 29
Description: The worst post-baseline score (lower scores are worse) through Day 29 in the clinical severity status 8-point ordinal scale, derived from all scores recorded after baseline up to and including Day 29. Participants with a score of 7 discharged to hospice care are considered as having a score of 1 (death) instead of a score of 7 for this endpoint.
  The clinical severity status 8-point ordinal scale scores are:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
  3. Hospitalized, on noninvasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities
Time Frame: Day 2 to Day 29
Population: Apremilast sub-protocol full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast + Standard of Care | Apremilast Placebo Control
Number analyzed (Participants) | 194 | 190
Participants
  1 (Death or discharged to hospice care) | 34 | 31
  2 (Hospitalized on invasive mechanical ventilation or ECMO) | 13 | 10
  3 (Hospitalized on noninvasive ventilation or high-flow oxygen devices) | 37 | 43
  4 (Hospitalized, requiring supplemental oxygen) | 75 | 62
  5 (Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care) | 21 | 35
  6 (Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care) | 0 | 0
  7 (Not hospitalized, limitation on activities and/or requiring home oxygen) | 5 | 2
  8 (Not hospitalized, no limitations on activities) | 5 | 5
  Missing | 4 | 2
Statistical Analysis 1: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Test type: Other; p = 0.4507, Proportional odds model; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.80 to 1.66] — [estimate comment as in outcome 17, analysis 1]

19. Secondary Outcome: Apremilast Sub-protocol: Number of Intensive Care Unit (ICU) Days From Day 1 Through Day 29
Description: as for outcome 9
Time Frame: Day 1 to Day 29
Population: Apremilast sub-protocol full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast + Standard of Care | Apremilast Placebo Control
Number analyzed (Participants) | 194 | 190
Participants
  0 days | 124 | 122
  1 day | 4 | 2
  2 days | 2 | 1
  3 days | 2 | 4
  4 days | 0 | 1
  5 days | 4 | 1
  6 days | 2 | 3
  7 days | 4 | 2
  8 days | 2 | 4
  9 days | 1 | 1
  10 days | 1 | 1
  11 days | 0 | 1
  12 days | 1 | 1
  13 days | 0 | 2
  14 days | 2 | 0
  15 days | 0 | 1
  17 days | 0 | 2
  18 days | 0 | 1
  20 days | 0 | 1
  21 days | 0 | 2
  23 days | 0 | 2
  25 days | 1 | 0
  27 days | 1 | 1
  28 days | 1 | 0
  29 days | 8 | 2
  30 days (death or discharged to hospice care) | 34 | 32
Statistical Analysis 1: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Test type: Other; p = 0.9741, Proportional odds model; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.64 to 1.53] — [estimate comment as in outcome 17, analysis 1]

20. Secondary Outcome: Apremilast Sub-protocol: Number of Invasive Mechanical Ventilator Days From Day 1 Through Day 29
Description: as for outcome 10
Time Frame: Day 1 to Day 29
Population: Apremilast sub-protocol full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast + Standard of Care | Apremilast Placebo Control
Number analyzed (Participants) | 194 | 190
Participants
  0 days | 147 | 147
  6 days | 1 | 1
  9 days | 1 | 0
  10 days | 1 | 0
  11 days | 1 | 1
  12 days | 0 | 1
  13 days | 2 | 0
  16 days | 0 | 2
  18 days | 0 | 1
  19 days | 1 | 0
  22 days | 1 | 0
  23 days | 0 | 1
  24 days | 0 | 1
  25 days | 3 | 1
  26 days | 1 | 1
  29 days | 1 | 0
  30 days (death or discharged to hospice care) | 34 | 33
Statistical Analysis 1: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Test type: Other; p = 0.8754, Proportional odds model; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.64 to 1.70] — [estimate comment as in outcome 17, analysis 1]

21. Secondary Outcome: Apremilast Sub-protocol: Percentage of Participants Who Achieved Clinical Recovery at Days 8, 15, and 29
Description: as for outcome 11
Time Frame: Day 8, Day 15, and Day 29
Population: Apremilast sub-protocol full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast + Standard of Care | Apremilast Placebo Control
Number analyzed (Participants) | 194 | 190
percentage of participants
  Day 8 | 36.6 | 35.8
  Day 15 | 57.7 | 60.0
  Day 29 | 66.0 | 72.1
Statistical Analysis 1: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Analysis of clinical recovery on Day 8; Test type: Other; p = 0.9695, Regression, Logistic; Risk Difference (RD) = 0.2, 95% CI 2-sided [-8.7 to 9.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Analysis of clinical recovery on Day 8; Test type: Other; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.64 to 1.59] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 3: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Analysis of clinical recovery on Day 15; Test type: Other; p = 0.6236, Regression, Logistic; Risk Difference (RD) = -2.4, 95% CI 2-sided [-11.9 to 7.1] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 4: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Analysis of clinical recovery on Day 15; Test type: Other; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.59 to 1.37] — [estimate comment as in outcome 14, analysis 2]
Statistical Analysis 5: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Analysis of clinical recovery on Day 29; Test type: Other; p = 0.1664, Regression, Logistic; Risk Difference (RD) = -6.2, 95% CI 2-sided [-14.9 to 2.5] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 6: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Analysis of clinical recovery on Day 29; Test type: Other; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.45 to 1.15] — [estimate comment as in outcome 14, analysis 2]

22. Secondary Outcome: Apremilast Sub-protocol: Percentage of Participants Who Achieved Sustained Clinical Recovery
Description: as for outcome 12
Time Frame: Day 60
Population: Apremilast sub-protocol full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Apremilast + Standard of Care | Apremilast Placebo Control
Number analyzed (Participants) | 194 | 190
percentage of participants | 66.0 | 66.3
Statistical Analysis 1: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Test type: Other; p = 0.9043, Regression, Logistic; Risk Difference (RD) = -0.5, 95% CI 2-sided [-9.3 to 8.3] — [estimate comment as in outcome 14, analysis 1]
Statistical Analysis 2: Comparison: Apremilast + Standard of Care vs Apremilast Placebo Control; Test type: Other; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.62 to 1.54] — [estimate comment as in outcome 14, analysis 2]

23. Secondary Outcome: Apremilast Sub-protocol: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to study treatment. A TEAE is an AE that occurs after the first dose of study drug. A serious AE is any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of hospitalization, resulted in persistent disability/incapacity, a congenital anomaly/birth defect, or an important medical event that may jeopardize the patient or require intervention to prevent an outcome listed above.
  The Investigator assessed the intensity of each AE according to the CTCAE grades:
  * Grade 1 Mild; asymptomatic or mild symptoms;
  * Grade 2 Moderate; minimal, local or noninvasive intervention indicated;
  * Grade 3 Severe or medically significant, not immediately life-threatening;
  * Grade 4 Life-threatening; urgent intervention indicated;
  * Grade 5 Death due to AE.
Time Frame: From first dose of study drug to end of study (Day 60)
Population: Apremilast safety analysis set included all participants in the apremilast FAS who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Apremilast + Standard of Care: Participants received 30 mg apremilast orally twice a day in addition to standard of care treatment for 14 days or until hospital discharge, whichever occurred first.
- Apremilast Placebo Control: Includes participants who received matching placebo to apremilast plus standard of care treatment as well as participants who received placebo to lanadelumab or placebo to zilucoplan plus standard of care treatment at a site concurrently enrolling apremilast sub-protocol participants and who would have been eligible for the apremilast sub-protocol.
- Apremilast Placebo + Standard of Care: Participants received matching placebo to apremilast orally twice a day in addition to standard of care treatment for 14 days or until hospital discharge, whichever occurred first.
Arm/Group | Apremilast + Standard of Care | Apremilast Placebo Control | Apremilast Placebo + Standard of Care
Number analyzed (Participants) | 189 | 187 | 182
Participants
  Any treatment-emergent adverse event (TEAE) | 102 | 103 | 100
  TEAE with a CTCAE grade ≥ 3 | 48 | 57 | 54
  Serious TEAE | 51 | 57 | 55
  TEAE leading to dose modification | 16 | 6 | 6
  TEAE leading to discontinuation of study drug | 9 | 12 | 11

24. Secondary Outcome: Zilucoplan Sub-protocol: Percentage of Participants Who Achieved Oxygen-Free Recovery at Day 29
Description: as for outcome 4
Time Frame: Day 29
Population: Zilucoplan sub-protocol full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zilucoplan + Standard of Care | Zilucoplan Placebo Control
Number analyzed (Participants) | 100 | 75
percentage of participants | 54.0 [43.74 to 64.02] | 60.0 [48.04 to 71.15]

25. Secondary Outcome: Zilucoplan Sub-protocol: Percentage of Participants With a ≥ 2-point Improvement From Baseline or Fit for Discharge on the Clinical Severity Status 8-Point Ordinal Scale at Day 29
Description: as for outcome 15
Time Frame: Baseline (Day 1) and Day 29
Population: Zilucoplan sub-protocol full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zilucoplan + Standard of Care | Zilucoplan Placebo Control
Number analyzed (Participants) | 100 | 7
percentage of participants | 66.0 [55.85 to 75.18] | 69.3 [57.62 to 79.47]

26. Secondary Outcome: Zilucoplan Sub-protocol: Percentage of Participants Who Died Before or on Day 29
Description: as for outcome 6
Time Frame: Day 1 to Day 29
Population: Zilucoplan sub-protocol full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zilucoplan + Standard of Care | Zilucoplan Placebo Control
Number analyzed (Participants) | 100 | 75
percentage of participants | 18.0 [11.03 to 26.95] | 24.0 [14.89 to 35.25]

27. Secondary Outcome: Zilucoplan Sub-protocol: Clinical Severity Status 8-Point Ordinal Scale Score at Days 8, 15, and 29
Description: The clinical severity status 8-point ordinal scale scores are:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or ECMO
  3. Hospitalized, on noninvasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities
  Participants with a score of 7 who were discharged to hospice care are counted with participants with a score of 1 (death) for this endpoint.
Time Frame: Day 8, Day 15, and Day 29
Population: Zilucoplan sub-protocol full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Zilucoplan + Standard of Care | Zilucoplan Placebo Control
Number analyzed (Participants) | 100 | 75
Participants
  Day 8: 1 (Death or discharged to hospice care) | 5 | 5
  Day 8: 2 (Hospitalized on invasive mechanical ventilation or ECMO) | 24 | 14
  Day 8: 3 (Hospitalized on noninvasive ventilation or high-flow oxygen devices) | 12 | 8
  Day 8: 4 (Hospitalized, requiring supplemental oxygen) | 16 | 14
  Day 8: 5 (Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care) | 5 | 10
  Day 8: 6 (Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care) | 0 | 1
  Day 8: 7 (Not hospitalized, limitation on activities and/or requiring home oxygen) | 22 | 9
  Day 8: 8 (Not hospitalized, no limitations on activities) | 11 | 12
  Day 8: Missing | 5 | 2
  Day 15: 1 (Death or discharged to hospice care) | 8 | 14
  Day 15: 2 (Hospitalized on invasive mechanical ventilation or ECMO) | 16 | 7
  Day 15: 3 (Hospitalized on noninvasive ventilation or high-flow oxygen devices) | 3 | 3
  Day 15: 4 (Hospitalized, requiring supplemental oxygen) | 10 | 6
  Day 15: 5 (Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care) | 2 | 2
  Day 15: 6 (Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care) | 0 | 1
  Day 15: 7 (Not hospitalized, limitation on activities and/or requiring home oxygen) | 25 | 14
  Day 15: 8 (Not hospitalized, no limitations on activities) | 31 | 26
  Day 15: Missing | 5 | 2
  Day 29: 1 (Death or discharged to hospice care) | 14 | 18
  Day 29: 2 (Hospitalized on invasive mechanical ventilation or ECMO) | 10 | 2
  Day 29: 3 (Hospitalized on noninvasive ventilation or high-flow oxygen devices) | 1 | 1
  Day 29: 4 (Hospitalized, requiring supplemental oxygen) | 5 | 1
  Day 29: 5 (Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care) | 1 | 0
  Day 29: 6 (Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care) | 0 | 2
  Day 29: 7 (Not hospitalized, limitation on activities and/or requiring home oxygen) | 20 | 14
  Day 29: 8 (Not hospitalized, no limitations on activities) | 44 | 35
  Day 29: Missing | 5 | 2

28. Secondary Outcome: Zilucoplan Sub-protocol: Worst Post-Baseline Score on Clinical Severity Status 8-Point Ordinal Scale From Baseline to Day 29
Description: The worst post-baseline score (lower scores are worse) through Day 29 in the clinical severity status 8-point ordinal scale scores, derived from all scores recorded after baseline up to and including Day 29. Participants with a score of 7 discharged to hospice care were considered as having a score of 1 (death) instead of a score of 7 for this endpoint.
  The clinical severity status 8-point ordinal scale scores scores are:
  1. Death
  2. Hospitalized, on invasive mechanical ventilation or ECMO
  3. Hospitalized, on noninvasive ventilation or high flow oxygen devices
  4. Hospitalized, requiring supplemental oxygen
  5. Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care
  7. Not hospitalized, limitation on activities and/or requiring home oxygen
  8. Not hospitalized, no limitations on activities
Time Frame: Day 2 to Day 29
Population: Zilucoplan sub-protocol full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Zilucoplan + Standard of Care | Zilucoplan Placebo Control
Number analyzed (Participants) | 100 | 75
Participants
  1 (Death or discharged to hospice care) | 14 | 18
  2 (Hospitalized on invasive mechanical ventilation or ECMO) | 21 | 6
  3 (Hospitalized on noninvasive ventilation or high-flow oxygen devices) | 24 | 12
  4 (Hospitalized, requiring supplemental oxygen) | 30 | 29
  5 (Hospitalized, not requiring supplemental oxygen, requiring ongoing medical care) | 5 | 7
  6 (Hospitalized, not requiring supplemental oxygen, no longer requires ongoing medical care) | 0 | 0
  7 (Not hospitalized, limitation on activities and/or requiring home oxygen) | 1 | 0
  8 (Not hospitalized, no limitations on activities) | 0 | 1
  Missing | 5 | 2

29. Secondary Outcome: Zilucoplan Sub-protocol: Number of Intensive Care Unit (ICU) Days From Day 1 Through Day 29
Description: as for outcome 9
Time Frame: Day 1 to Day 29
Population: Zilucoplan sub-protocol full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Zilucoplan + Standard of Care | Zilucoplan Placebo Control
Number analyzed (Participants) | 100 | 75
Participants
  0 days | 56 | 34
  1 day | 0 | 2
  3 days | 2 | 2
  4 days | 0 | 1
  5 days | 1 | 1
  6 days | 1 | 3
  7 days | 4 | 0
  8 days | 0 | 4
  9 days | 3 | 1
  10 days | 0 | 1
  11 days | 1 | 0
  13 days | 1 | 2
  14 days | 1 | 0
  15 days | 0 | 1
  17 days | 1 | 1
  18 days | 1 | 0
  21 days | 0 | 2
  22 days | 1 | 0
  25 days | 1 | 0
  26 days | 1 | 0
  29 days | 8 | 2
  30 days (death or discharged to hospice care) | 17 | 18

30. Secondary Outcome: Zilucoplan Sub-protocol: Number of Invasive Mechanical Ventilator Days From Day 1 Through Day 29
Description: as for outcome 10
Time Frame: Day 1 to Day 29
Population: Zilucoplan sub-protocol full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Zilucoplan + Standard of Care | Zilucoplan Placebo Control
Number analyzed (Participants) | 100 | 75
Participants
  0 days | 67 | 52
  6 days | 0 | 1
  7 days | 4 | 0
  9 days | 1 | 0
  10 days | 1 | 0
  12 days | 0 | 1
  13 days | 1 | 0
  16 days | 0 | 1
  18 days | 1 | 0
  22 days | 1 | 0
  24 days | 1 | 1
  25 days | 1 | 0
  26 days | 1 | 1
  27 days | 1 | 0
  28 days | 1 | 0
  29 days | 1 | 0
  30 days (death or discharged to hospice care) | 18 | 18

31. Secondary Outcome: Zilucoplan Sub-protocol: Percentage of Participants Who Achieved Clinical Recovery by Days 8, 15, and 29
Description: as for outcome 11
Time Frame: Day 8, Day 15, and Day 29
Population: Zilucoplan sub-protocol full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zilucoplan + Standard of Care | Zilucoplan Placebo Control
Number analyzed (Participants) | 100 | 75
percentage of participants
  Day 8 | 33.0 [23.92 to 43.12] | 30.7 [20.53 to 42.38]
  Day 15 | 53.0 [42.76 to 63.06] | 53.3 [41.45 to 64.95]
  Day 29 | 60.0 [49.72 to 69.67] | 66.7 [54.83 to 77.14]

32. Secondary Outcome: Zilucoplan Sub-protocol: Percentage of Participants Who Achieved Sustained Clinical Recovery
Description: as for outcome 12
Time Frame: Day 60
Population: Zilucoplan sub-protocol full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Zilucoplan + Standard of Care | Zilucoplan Placebo Control
Number analyzed (Participants) | 100 | 75
percentage of participants | 55.0 [44.73 to 64.97] | 64.0 [52.09 to 74.77]

33. Secondary Outcome: Zilucoplan Sub-protocol: Number of Participants With Treatment-emergent Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to study treatment. A TEAE is an AE that occurs after the first dose of study drug. A serious AE is any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of hospitalization, resulted in persistent disability/incapacity, a congenital anomaly/birth defect, or an important medical event that may jeopardize the patient or require intervention to prevent an outcome listed above.
  The Investigator assessed the intensity of each AE according to the CTCAE grades:
  * Grade 1 Mild; asymptomatic or mild symptoms;
  * Grade 2 Moderate; minimal, local or noninvasive intervention indicated;
  * Grade 3 Severe or medically significant, not immediately life-threatening;
  * Grade 4 Life-threatening; urgent intervention indicated;
  * Grade 5 Death due to AE.
Time Frame: From first dose of study drug to end of study (Day 60)
Population: Zilucoplan safety analysis set included all participants in the zilucoplan FAS who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Zilucoplan+ Standard of Care: Participants received 32.4 mg zilucoplan by subcutaneous injection every day for 14 days, or until discharge if discharge was before 14 days of treatment, in addition to standard of care.
- Zilucoplan Placebo Control: Includes participants who received matching placebo to zilucoplan plus standard of care treatment as well as participants who received placebo to lanadelumab or placebo to apremilast plus standard of care treatment at a site that enrolled at least one participant in the zilucoplan sub-protocol.
- Zilucoplan Placebo + Standard of Care: Participants received placebo to zilucoplan by subcutaneous injection every day for 14 days, or until discharge if discharge was before 14 days of treatment, in addition to standard of care.
Arm/Group | Zilucoplan+ Standard of Care | Zilucoplan Placebo Control | Zilucoplan Placebo + Standard of Care
Number analyzed (Participants) | 95 | 73 | 7
Participants
  Any treatment-emergent adverse event (TEAE) | 65 | 47 | 4
  TEAE with a CTCAE grade ≥ 3 | 34 | 29 | 3
  Serious TEAE | 31 | 29 | 2
  TEAE leading to dose modification | 0 | 5 | 0
  TEAE leading to discontinuation of study drug | 7 | 5 | 1

ADVERSE EVENTS:
Time Frame: From first dose of study drug to end of study (Day 60).
Description: All-cause mortality is reported for all randomized participants, according to randomized treatment group.
  Adverse events are reported for all participants who received at least one dose of study drug, according to study drug received.
Groups:
- Lanadelumab + SoC: Participants received lanadelumab 300 mg by intravenous infusion on Day 1, and a second dose administered on Day 4, in addition to standard of care (SoC).
- Lanadelumab Placebo + SoC: Participants received placebo to lanadelumab by intravenous infusion on Day 1, and a second dose administered on Day 4 in, addition to standard of care.
- Apremilast + SoC: Participants received 30 mg apremilast orally twice a day in addition to standard of care treatment for 14 days or until hospital discharge, whichever occurred first.
- Apremilast Placebo + SoC: Participants received matching placebo to apremilast orally twice a day in addition to standard of care treatment for 14 days or until hospital discharge, whichever occurred first.
- Zilucoplan + SoC: Participants received 32.4 mg zilucoplan by subcutaneous injection every day for 14 days, or until discharge if discharge was before 14 days of treatment, in addition to standard of care.
- Zilucoplan Placebo + SoC: Participants received placebo to zilucoplan by subcutaneous injection every day for 14 days, or until discharge if discharge was before 14 days of treatment, in addition to standard of care.
Arm/Group | Lanadelumab + SoC | Lanadelumab Placebo + SoC | Apremilast + SoC | Apremilast Placebo + SoC | Zilucoplan + SoC | Zilucoplan Placebo + SoC
All-Cause Mortality (participants affected / at risk) | 8/28 | 1/1 | 37/194 | 35/184 | 20/100 | 3/8
Serious Adverse Events (participants affected / at risk) | 11/27 | 1/1 | 51/189 | 55/182 | 31/95 | 2/7
Other Adverse Events (participants affected / at risk) | 12/27 | 1/1 | 63/189 | 50/182 | 46/95 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lanadelumab + SoC (N=27) | Lanadelumab Placebo + SoC (N=1) | Apremilast + SoC (N=189) | Apremilast Placebo + SoC (N=182) | Zilucoplan + SoC (N=95) | Zilucoplan Placebo + SoC (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 2 | 3 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 2 | 2 | 2 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiovascular insufficiency (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Blindness unilateral (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 3 | 2 | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 5 | 2 | 0
COVID-19 pneumonia (Infections and infestations) | 3 | 1 | 6 | 6 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Nosocomial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 4 | 3 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 1 | 1 | 2 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 3 | 3 | 1 | 0
Septic shock (Infections and infestations) | 2 | 0 | 12 | 10 | 8 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Procedural shock (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Propofol infusion syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Coma (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 7 | 4 | 7 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 4 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 11 | 6 | 5 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3 | 2 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6 | 5 | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 14 | 10 | 8 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
Haemodynamic instability (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lanadelumab + SoC (N=27) | Lanadelumab Placebo + SoC (N=1) | Apremilast + SoC (N=189) | Apremilast Placebo + SoC (N=182) | Zilucoplan + SoC (N=95) | Zilucoplan Placebo + SoC (N=7)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 9 | 4 | 9 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 5 | 4 | 3 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 1 | 3 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 3 | 2 | 4 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 9 | 10 | 16 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 9 | 5 | 3 | 0
Pyrexia (General disorders) | 3 | 0 | 4 | 6 | 9 | 1
Bacterial infection (Infections and infestations) | 1 | 0 | 4 | 1 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 5 | 0 | 3 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1 | 0 | 2 | 2 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 4 | 2 | 5 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Procalcitonin increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 4 | 3 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 8 | 7 | 3 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 1 | 4 | 3 | 3 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 4 | 6 | 5 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 8 | 3 | 8 | 0
Headache (Nervous system disorders) | 0 | 0 | 10 | 3 | 2 | 0
Depression (Psychiatric disorders) | 2 | 0 | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 8 | 5 | 8 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 1 | 11 | 5 | 2 | 1
Oliguria (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 5 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 3 | 2 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1 | 3 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 3 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 3 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 4 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 8 | 7 | 10 | 0
Hypotension (Vascular disorders) | 1 | 0 | 5 | 9 | 13 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT04590586/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/86/NCT04590586/SAP_001.pdf